CLINICAL TRIAL: NCT00416221
Title: Development and a Pilot Study of the PACEPRO Exercise and Mood Management Program in Depressed Patients on Escitalopram Oxalate (Lexapro)
Brief Title: PACEPro - Mood Management Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Forest Laboratories (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LXP-MD-106; 2005-3889(UCSD Number)
Record Dates: First submitted 2006-12-22; First posted 2006-12-27 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Depression
Keywords: Depression; Lexapro
MeSH Terms: conditions — Depression | interventions — Escitalopram; Exercise

INTERVENTIONS:
Drug: Lexapro, an antidepressant medicine
Behavioral: Physical Activity
Behavioral: Mood Management Skills
Behavioral: Personalized support from a Family Nurse Practitioner

SUMMARY:
Researchers at the University of California at San Diego (UCSD) are conducting a 12-week study to test the PACEPRO program. This program is designed to reduce depression by providing:

Lexapro, an antidepressant medicine…Learn More Physical activity information and pedometer Mood management skills and a Mood Mastery Guide Personalized support from a Family Nurse Practitioner

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with mild to moderate depression
* Are willing to take the antidepressant Lexapro
* Can access and use Email and the Internet
* Are willing and able to be physically active
* Access to a primary care physician

Exclusion Criteria:

Subjects will be excluded from participation for the following reasons:

* Pregnancy or breastfeeding
* Narrow angle glaucoma
* Any uncontrolled medical condition or any medical condition which would represent a contraindication to Escitalopram Oxalate Lexapro® pharmacotherapy. Any concomitant non-psychotropic medications that the physician determines are a contraindication to Escitalopram Oxalate Lexapro® pharmacotherapy Bipolar disorder, or any psychotic or organic mental disorder or dementia
* History of intolerance or allergy to Lexapro, or of prior failed treatment for depression with Lexapro
* Current substance abuse or dependency
* Current active suicidal ideation
* Current use of herbal psychoactive treatments such as St. John's Wort
* Concurrent psychotropic medication is not permitted for 2 weeks prior to randomization (4 weeks in the case of fluoxetine) or at any point after
* Receipt of formal psychotherapy concurrently
* Inability, in the investigator's opinion, to comply with study procedures or assessments
* Inability to exercise

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Measurement visits will be conducted at the PACE office. The specific activities to be conducted at the baseline, 6 and 12 week assessment visits are listed below.
Physiological Measures | baseline, 6 weeks, 12 weeks
Height and weight | baseline, 6 weeks, 12 weeks
Waist & hip, circumference | baseline, 6 weeks, 12 weeks
Blood pressure and pulse | baseline, 6 weeks, 12 weeks
Physical activity level measured by wearing a monitor around the waist for 3 days (at baseline and 12 weeks only) | baseline, 6 weeks, 12 weeks
Interview/Survey Measures | baseline, 6 weeks, 12 weeks
Self report depressive symptoms | baseline, 6 weeks, 12 weeks
Self-report of moderate and vigorous physical activity for seven days | baseline, 6 weeks, 12 weeks
Self-report of TV viewing and recreational computer use for seven days | baseline, 6 weeks, 12 weeks
Self-report on readiness to make changes in physical activity and mood management behaviors | baseline, 6 weeks, 12 weeks
Personal assessment of factors related to behavior change including: self-efficacy, social support, barriers to change, and use of behavior change skills, and the environment | baseline, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Patrick, MD, MS, Principal Investigator — UCSD; Catherine Pearson-Bennett, MSN, RN, Study Director — UCSD
Locations (1):
- UCSD Professional Building, La Jolla, California, United States